CLINICAL TRIAL: NCT05074485
Title: Discovery and Analytical Validation of Inflammatory Bio-signatures of the Human Pain Experience
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alan Prossin (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Alan Prossin, Assistant Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-19-0627; R61NS113316 (NIH)
Record Dates: First submitted 2021-09-27; First posted 2021-10-12 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo plus nociceptive pain challenge, then anakinra plus nociceptive pain challenge (Experimental): Pharmacological challenge (with placebo) plus nociceptive pain challenge, then pharmacological challenge (with anakinra) plus nociceptive pain challenge
  Interventions: Drug: anakinra; Drug: Placebo; Other: Nociceptive pain challenge
- Anakinra plus nociceptive pain challenge, then placebo plus nociceptive pain challenge (Experimental): Pharmacological challenge (with anakinra) plus nociceptive pain challenge, then pharmacological challenge (with placebo) plus nociceptive pain challenge
  Interventions: Drug: anakinra; Drug: Placebo; Other: Nociceptive pain challenge

INTERVENTIONS:
Drug: anakinra — intravenous injection of 100 milligrams anakinra
  Other Names: Kineret
Drug: Placebo — intravenous injection of 1 milliliter normal saline
  Other Names: Inert Substance
Other: Nociceptive pain challenge — The experimental, standardized, nociceptive pain challenge will induce a moderate level of sustained pain. The pain challenge involves a masseteric injection in the left or right jaw muscle of normal saline (0.15 ml bolus of 0.9% normal saline) over a 15 second period followed by continuous infusion via a closed loop infusion system for 20 minutes.
  Other Names: Pain Induction

SUMMARY:
The first objective of the study is to evaluate whether a novel bio-signature (derived from a wide range of pro- and anti-nociceptive IL-1 family cytokine activity) will predict pain experienced and also release of underlying endogenous opioid neurotransmitters during an experimental nociceptive pain challenge, which will be performed while simultaneously quantifying mu-opioid receptor activity in the brain via [11C]-carfentanil PET neuroimaging in healthy subjects. Another objective is to evaluate whether an anti-inflammatory drug that reduces activation of IL-1b (minocycline) will perturb the balance between pro- and anti-nociceptive IL-1 cytokines and effect a reduction in pain experienced (and endogenous opioids released) during the experimental, nociceptive pain challenge. A final objective is to evaluate performance characteristics (sensitivity, accuracy, dynamic range) of the biosignature for the purpose of predicting post-operative pain.

DETAILED DESCRIPTION:
Lack of precision in tools that quantify risk and assess presentation of post-operative pain poses substantial burden to prevention and treatment and is a major contributor to the nationwide opioid epidemic. Enhanced precision in post- operative pain care requires quantitative tools that individualize assessment of widely variant human pain experiences, accounting for variance in intensity, threshold, and in both affective and sensory components of pain. No currently available measure is sufficiently sensitive, accurate, and reliable to account for the wide variance in risk or clinical presentation of post-operative pain that is required to impact best practices. To address this unmet need, we will discover (R61 phase) and validate (R33 phase) a novel, fit-for-purpose, objective bio-signature that is sensitive, accurate, and reliable in predicting risk (and presentation) of post-operative pain states following a elective cosmetic surgery (e.g. abdominoplasty), a body contouring surgery frequently performed and associated with post-operative pain.

Evidence suggests it is biologically plausible to develop a bio-signature of the human pain experience that derives from IL-1 family cytokine activity. In animal models, imbalance between pro- and anti-nociceptive IL-1 family cytokines is readily induced pharmacologically and surgically, enhancing pain behavior, central endogenous opioid release, and tolerance to opioid analgesics, all factors that contribute to chronicity. Pharmacologic blockade of pro-nociceptive IL-1 cytokines with soluble IL-1ra reverses the pro-nociceptive effects. Evidence suggests similar relationships exist in humans. Concentration of IL-1b sampled intra-operatively from wound site blood revealed predicts surgical complications and post-operative pain. However, IL-1b (on its own) has not proven sufficiently accurate, sensitive, or reliable to account for the broad inter-individual variance in risk and clinical presentation of human post-operative pain states. In preliminary data from separate regression analyses, neither IL-1b nor IL-1ra significantly predicted pain (intensity or threshold). However, regression models incorporating both IL-1b and IL-1ra showed that imbalance between these 2 factors (pro-nociceptive IL-1bias) synergistically enhanced prediction of pain (intensity and threshold) and underlying endogenous opioid release during a standardized pain challenge, accounting for 20% of the pain variance. IL-1b (pro-nociceptive) was a positive predictor and IL-1ra (anti-nociceptive) a negative predictor of pain. Including additional variance factors (sex, mu-opioid receptor polymorphism, neuroticism) in the model accounted for another 5% of the pain variance. Pain variance factors can impact concentration of additional IL-1 cytokines that regulate IL-1 signaling, suggesting it is both biologically and statistically plausible that incorporating a wide array of IL-1 family cytokines (IL-1b, IL-1ra, IL-1a, sIL-1r1, IL-1RAcP, IL-18, IL-18bp, IL-18Ra, IL-18Rb, IL-36, IL-38, IL-33, sTLR4) into a broader bio-signature of IL-1 family cytokine activity will perform superior to simple measures of IL-1bias (that include only IL-1b and IL-1ra) in predicting the highly heterogeneous human post-operative pain experience.

This study phase focuses on discovery (and analytic validation) of a novel, bio-signature of risk for post-operative pain states and underlying opioid-cytokine interactions. Performance (accuracy, sensitivity, dynamic range) in predicting experimental and post-operative pain will be tested in n=70 healthy humans following elective abdominoplasty.

More Specifically, The first objective of the study is to evaluate whether a novel bio-signature (derived from a wide range of pro- and anti-nociceptive IL-1 family cytokine activity) will predict pain experienced and also release of underlying endogenous opioid neurotransmitters during an experimental nociceptive pain challenge, which will be performed while simultaneously quantifying mu-opioid receptor activity in the brain via [11C]-carfentanil PET neuroimaging in healthy subjects. Another objective is to evaluate whether an anti-inflammatory drug that reduces activation of IL-1b (anakinra) will perturb the balance between pro- and anti-nociceptive IL-1 cytokines and effect a reduction in pain experienced (and endogenous opioids released) during the experimental, nociceptive pain challenge. A final objective is to evaluate performance characteristics (sensitivity, accuracy, dynamic range) of the biosignature for the purpose of predicting post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Obese or non-obese
* Awaiting elective surgery
* Negative urine pregnancy test

Exclusion Criteria:

* Active, severe medical or psychiatric illness (per DSM-V)
* History of depressive and/or anxiety symptoms with or without presence of a DSM-V depressive and/or anxiety disorder
* Current or recent (within past 3 months) suicidal thoughts/plans/attempts
* Current or recent (within past 3 months) substance use/abuse/dependence (Note: stable nicotine use is acceptable, non-risky alcohol use is acceptable)
* Active or chronic medical illness (except obesity: either obese or non-obese volunteers can enroll in the study).
* MRI exclusion criteria including presence of non-MRI-safe medical device(s), magnetizable objects in soft tissue, severe claustrophobia, etc.
* Recent (past year) PET scan(s).
* Lifetime excessive radiation exposure that would be exclusionary via standards of the local radiation safety committee.
* Current medication treatment that would impact measures of interest.
* Current pregnancy or recent (within the past 2 months) intercourse without an acceptable contraceptive method
* Exclusion criteria for Anakinra treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Pain as assessed by total pain score on the McGill Pain Questionnaire | 0 minutes, This represents the study baseline, prior to any brain imaging
  The total pain score on the McGill Pain Questionnaire ranges from 0-78, with a higher score indicating greater pain.
Pain as assessed by total pain score on the McGill Pain Questionnaire | 90 minutes, upon completion of brain imaging
  The total pain score on the McGill Pain Questionnaire ranges from 0-78, with a higher score indicating greater pain.
Pain as assessed by total pain score on the McGill Pain Questionnaire | 12 to 24 hours before elective surgery
  The total pain score on the McGill Pain Questionnaire ranges from 0-78, with a higher score indicating greater pain.
Pain as assessed by total pain score on the McGill Pain Questionnaire | 24 to 48 hours after elective surgery
  The total pain score on the McGill Pain Questionnaire ranges from 0-78, with a higher score indicating greater pain.
Pain as assessed by total pain score on the McGill Pain Questionnaire | 6 to 8 weeks after elective surgery
  The total pain score on the McGill Pain Questionnaire ranges from 0-78, with a higher score indicating greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Prossin, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No